CLINICAL TRIAL: NCT07245355
Title: Effects of Recreational Exercises (Swimming, Pilates, and Walking) on Muscle Strength and Balance in Women at Risk for Osteoporosis
Brief Title: Contribution of Recreational Exercises to Balance and Muscle Strength in Osteoporosis Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Nur ALP, Lecturer, MSc., Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SuleymanDU-97/14
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis (Senile)
Keywords: osteoporosis; Recreational Exercise
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: The study is planned as a randomized controlled prospective trial. Participants were assigned to three groups using a computer-generated random number table (n=20).
  Pilates Group: Mat Pilates was performed three days a week for 45 minutes. Swimming Group: Moderate-intensity swimming was performed 3 days a week for 40 minutes.
  Walking Group: Brisk walking was performed 3 days a week for 45 minutes.
Who Masked: Participant
Masking Description: A single-blind study was designed in which the patients would be unaware of their group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates Group (Experimental): Pilates Group: Mat Pilates was performed three days a week for 45 minutes. The programme included a 10-minute warm-up, 30 minutes of basic Pilates exercises (hundred, roll-up, spine stretch, single leg stretch) and a 5-minute cool-down and stretching phase. The exercises were conducted by a certified Pilates instructor.
  Interventions: Other: Experimental Group 1
- Swimming Group (Experimental): Swimming Group: Moderate-intensity swimming was performed 3 days a week for 40 minutes. The exercises included a 5-minute warm-up, 30 minutes of freestyle and backstroke swimming, and a 5-minute cool-down phase. Participants' heart rates were maintained at 60- 70% of their maximum heart rate.
  Interventions: Other: Experimental Group 2
- Walking Group (Experimental): Brisk walking was performed 3 days a week for 45 minutes. The programme consisted of a 5-minute warm-up walk, 35 minutes of walking at 60-70% of maximum heart rate, and a 5-minute cool-down walk.
  Interventions: Other: Experimental Group 3

INTERVENTIONS:
Other: Experimental Group 1 — Sixty women aged 40-60 years with a T-score between -1.0 and -2.5 were randomly assigned to three groups (Pilates, Swimming, Walking; n=20). Participants exercised for 40-45 minutes three days a week for 12 weeks.All exercises in this group were conducted by a certified Pilates instructor. Pilates exercises were performed on a mat.Session Content:
  Warm-Up (10 min): Breathing exercises, shoulder rotation, neck stretch, posterior pelvic tilt, and spinal mobilization exercises were performed.
  Main Section (30 min):
  Weeks 1-4: Basic movements - Hundred, Roll-Up, Single Leg Stretch, Spine Stretch Weeks 5-8: Intermediate variations - Double Leg Stretch, Rolling Like a Ball, Saw Weeks 9-12: Advanced balance-focused movements - Teaser Prep, Side Kick Series, Swimming, Leg Pull Front Cool-Down (5 min): Deep breathing exercises, hamstring stretching, and spinal Participation rates were regularly recorded, and individuals who participated below 80% of the program were excluded from the analysis.
  Arms: Pilates Group
Other: Experimental Group 2 — Participants in the swimming group completed moderate-intensity swimming exercises for 40 minutes, three days a week. The program consisted of a 5-minute warm-up, 30 minutes of freestyle and backstroke swimming, and a 5-minute cool-down. Participants' heart rates were maintained between 60 and 70% of their maximum heart rate.
  Session content:
  Warm-up (5 min): Light swimming, in-water mobilization exercises
  Main Part (30 min):
  Weeks 1-4: Freestyle swimming with 25-50 m rest intervals Weeks 5-8: Alternating freestyle and backstroke swimming with 75-100 m rest intervals.
  Weeks 9-12: Continuous swimming sets (150-200 m) - technical development and endurance Cool down (5 min): Light swimming, stretching in the water Exercise intensity was monitored using the Borg Scale of Perceived Exertion (RPE). Participation rates were regularly recorded, and individuals who participated below 80% of the program were excluded from the analysis.
  Arms: Swimming Group
Other: Experimental Group 3 — Individuals in this group participated in brisk walking at 60-70% of their maximum heart rate for 45 minutes, three days a week. The program consisted of a 5-minute warm-up walk, a 35-minute brisk walk, and a 5-minute cool-down walk. A 45-minute walking program was designed three days a week (Tuesday, Thursday, Saturday).
  Terrace: Flat, safe walking track Intensity: 60-70% of maximum heart rate
  Session Contents:
  Warm-Up (5 min): Light walking, shoulder and hip mobilization
  Main Part (35 min):
  Weeks 1-4: 5-6 km/h brisk walking Weeks 5-8: 6-6.5 km/h brisk walking Weeks 9-12: 6.5-7 km/h brisk walking Cool-Down (5 min): Slow walking, calf, hamstring, and lower back stretching exercises.Exercise intensity was monitored in all groups using the Borg Scale of Perceived Exertion (RPE). Participation rates were regularly recorded, and individuals who participated below 80% of the program were excluded from the analysis.
  Arms: Walking Group

SUMMARY:
This study aims to evaluate the effects of recreational exercises such as Pilates, swimming and walking on muscle strength and balance in women at risk of osteoporosis.

Study hypotheses:

H1: Pilates exercises will be more effective than walking exercises in improving muscle strength among women at risk of osteoporosis.

H2: Swimming exercises will be more effective than walking exercises in improving muscle strength among women at risk of osteoporosis.

H3: Pilates exercises will be more effective than walking exercises in improving balance among women at risk of osteoporosis.

H4: Swimming exercises will be more effective than walking exercises in improving balance among women at risk of osteoporosis.

H5: Pilates and swimming exercises will have similar effects on improving muscle strength and balance among women at risk of osteoporosis.

DETAILED DESCRIPTION:
Participants were selected from among women who had previously been diagnosed with osteoporosis risk by a physician and who applied to the Isparta Merwellness Pilates gym for exercise.

The study is planned as a randomized controlled prospective trial. Participants were assigned to three groups using a computer-generated random number table (n=20).

Pilates Group: Mat Pilates was performed three days a week for 45 minutes. Swimming Group: Moderate-intensity swimming was performed 3 days a week for 40 minutes.

Walking Group: Brisk walking was performed 3 days a week for 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Having a sedentary lifestyle (not having exercised regularly in the past 6 months),
2. No musculoskeletal or neurological conditions that would prevent participation,
3. Voluntarily agreeing to participate in the study.

Exclusion Criteria:

1. Use of medications affecting bone metabolism (e.g., bisphosphonates, corticosteroids),
2. History of fracture within the past 6 months,
3. Uncontrolled cardiovascular or metabolic diseases.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength | At baseline and at the end of the 12-week intervention
  Handgrip strength was measured using a digital hand dynamometer (Jamar Plus+, kg). Three repetitions were taken during the measurements, and the highest value was recorded. The Jamar dynamometer has high reliability in individuals with osteoporosis (ICC = 0.95).
Trunk flexor and extensor strength | At baseline and at the end of the 12-week intervention
  Trunk flexor and extensor strength were assessed using isokinetic dynamometry (Biodex System 4) at a speed of 60°/s. This method has been reported as a valid measurement tool for elderly individuals and those at risk of osteoporosis.
Berg Balance Scale (BBS) | At baseline and at the end of the 12-week intervention
  Berg Balance Scale (BBS): A 14-item test scored between 0 and 56. The reliability coefficient in the Turkish adaptation was found to be 0.98.
Computerised posturography: | At baseline and at the end of the 12-week intervention
  Computerised posturography: Static and dynamic balance were assessed, and centre of pressure (CoP) oscillation (mm) was recorded. Posturography is a widely used objective method in the osteoporotic population.

CONTACTS AND LOCATIONS:
Overall Officials: HULUSİ ALP, Professor, Study Director — Suleyman Demirel University
Locations (1):
- Süleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data for objectives of the research will be compared after they are received.